CLINICAL TRIAL: NCT00544713
Title: Evaluate the Safety and Efficacy of a New Artificial Tear for Use After LASIK Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AG9818-001
Record Dates: First submitted 2007-10-12; First posted 2007-10-16 (Estimated); Results first posted 2011-12-14 (Estimated); Last update posted 2011-12-14 (Estimated); Status verified 2011-11

CONDITIONS: Dry Eye Syndrome
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Carboxymethylcellulose Sodium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Carboxymethylcellulose and Glycerin based artificial tear (Experimental): Carboxymethylcellulose and Glycerin based artificial tear
  Interventions: Drug: Carboxymethylcellulose and Glycerin based artificial tear
- Carboxymethylcellulose based artificial tear (Active Comparator): Carboxymethylcellulose based artificial tear
  Interventions: Drug: Carboxymethylcellulose

INTERVENTIONS:
Drug: Carboxymethylcellulose and Glycerin based artificial tear — As directed by Investigator at the end of each study visit: 1 to 2 drops in each eye, 1 to 2 times a day up to every hour while awake
  Arms: Carboxymethylcellulose and Glycerin based artificial tear
Drug: Carboxymethylcellulose — As directed by Investigator at the end of each study visit: 1 to 2 drops in each eye, 1 to 2 times a day up to every hour while awake
  Other Names: Refresh Plus®
  Arms: Carboxymethylcellulose based artificial tear

SUMMARY:
This study will evaluate the safety and efficacy of a new artificial tear for the treatment of dry eye that may occur after LASIK surgery

ELIGIBILITY:
Inclusion Criteria:

* Candidate for bilateral LASIK surgery for myopia correction in the range of -1.00 to -8.00 diopters

Exclusion Criteria:

* Dry eye signs and symptoms
* Preoperative soft or rigid contact lens wear within last 7 or 30 days, respectively
* Pregnancy or planning pregnancy
* Uncontrolled systemic disease
* Use of systemic medications affecting dry eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2007-09; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Carboxymethylcellulose and Glycerin Based Artificial Tear | Carboxymethylcellulose Based Artificial Tear
Started | 114 | 114
Completed | 111 | 109
Not Completed | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Carboxymethylcellulose and Glycerin Based Artificial Tear | Carboxymethylcellulose Based Artificial Tear | Total
Number analyzed (Participants) | 114 | 114 | 228
Age, Customized [Number; unit: participants]
  <40 Years | 88 | 92 | 180
  >= 40 Years | 26 | 22 | 48
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 51 | 113
  Male | 52 | 63 | 115

OUTCOME MEASURES:

1. Primary Outcome: Post LASIK Dry Eye Symptoms as Measured by Ocular Surface Disease Index (OSDI©) Score at Day 90
Description: Measured on 12 domains (categories); a 5-point scale for each domain (0 = best, no dry eye symptoms, 4 = worst, constant dry eye symptoms). Sum of the domain scores is normalized (standardized) to a severity scale of 0-100 (0 = no symptoms (best score), 100 = maximum severity (worst score)).
Time Frame: Day 90
Population: Intent to Treat population defined as all patients who started the study and were randomized
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Carboxymethylcellulose and Glycerin Based Artificial Tear | Carboxymethylcellulose Based Artificial Tear
Number analyzed (Participants) | 114 | 114
Scores on a Scale | 8.32 (11.125) | 6.43 (8.036)

2. Secondary Outcome: Patient Acceptability- Percentage of Patients Who Rated Artificial Tears (AT) as Acceptable at Day 90
Description: A questionnaire was administered to all patients to evaluate the acceptability of the Artificial Tears (referred to as AT). Percentage of patients responding either "Agree" or "Strongly Agree" at day 90 was tabulated. The potential response categories included "Strongly Agree", "Agree", "Neither Agree Nor Disagree", "Disagree" and "Strongly Disagree".
Time Frame: Day 90
Population: Intent to Treat includes all patients who started the study are were randomized. Only those patients who answered the particular question on Day 90 were analyzed. This is indicated in parenthesis as (number of patients in the first arm who answered that specific question/Number of patients in the second arm who answered that specific question).
Measure: Number; unit: Percentage of Patients
Arm/Group | Carboxymethylcellulose and Glycerin Based Artificial Tear | Carboxymethylcellulose Based Artificial Tear
Number analyzed (Participants) | 114 | 114
Percentage of Patients
  Liked using these AT (112/110) | 88.4 | 93.6
  AT helped eyes feel comfortable (112/110) | 94.6 | 94.5
  AT were soothing to eyes (111/110) | 95.5 | 95.4
  AT protected eyes from dryness (112/109) | 88.4 | 89.9
  AT protected eyes from low humidity (112/110) | 78.6 | 82.7
  Vision was normal few min.after AT use(112/110) | 93.8 | 92.7
  Few min. after use, AT gave clear vision(111/110) | 94.6 | 94.5
  AT helped eyes heal from surgery (112/110) | 83.9 | 86.4
  AT helped eyes feel same as pre-LASIK (111/110) | 85.6 | 89.1
  It's good to use AT after surgery(111/109) | 97.3 | 96.3

3. Secondary Outcome: Patient Acceptability (Sensory) - Percentage of Patients Who Rated Artificial Tears (AT) as Acceptable at Day 90
Description: A patient acceptability - sensory questionnaire was administered to all patients to evaluate the acceptability of the Artificial Tears (AT). Percentage of patients responding either "Agree" or "Strongly Agree" at day 90 was tabulated. The potential response categories included "Strongly Agree", "Agree", "Neither Agree Nor Disagree", "Disagree" and "Strongly Disagree".
Time Frame: Day 90
Population: Intent to Treat includes all patients who started the study and were randomized. Only those patients who answered the particular question on Day 90 were analyzed. This is indicated in parenthesis as (number of patients in the first arm who answered that specific question/Number of patients in the second arm who answered that specific question).
Measure: Number; unit: Percentage of Patients
Arm/Group | Carboxymethylcellulose and Glycerin Based Artificial Tear | Carboxymethylcellulose Based Artificial Tear
Number analyzed (Participants) | 114 | 114
Percentage of Patients
  Thickness of AT is just right (112/109) | 79.5 | 87.2
  AT did not interfere with vision (112/108) | 64.3 | 82.4
  AT did not cause my eyes to get crusty (112/108) | 66.1 | 80.6
  AT were easy to use (112/109) | 99.1 | 99.1
  AT were convenient to use (112/109) | 96.4 | 91.7
  AT were important to a good outcome (111/109) | 82.0 | 80.7
  AT were helpful to achieve comfort (112/109) | 92.0 | 93.6
  AT were helpful to achieve good vision (112/109) | 71.4 | 76.1
  I no longer feel I need to use AT (111/108) | 43.2 | 38.0

4. Secondary Outcome: Best Corrected Visual Acuity (BCVA) Status at Day 90
Description: BCVA status at Day 90 reported as the number of patients whose scores were either "Better", "No Change", or "Worse" than their scores at baseline. The status was tabulated as number of lines read correctly at Day 90 minus the number of lines read correctly at baseline. "Better" equals increase of 2 lines or more; "No Change" equals change between -2 to +2 lines; "Worse" equals decrease of 2 lines or more. BCVA is measured using a special eye chart a nd is reported as the number of lines (5 letters per line) read correctly.
Time Frame: Day 90
Population: Intent to Treat includes all patients who started the study and were randomized. One patient's status in the first arm was not available at Day 90 and was not evaluated for this outcome measure therefore only 113 patients were analyzed for this outcome measure.
Measure: Number; unit: Number of Patients
Arm/Group | Carboxymethylcellulose and Glycerin Based Artificial Tear | Carboxymethylcellulose Based Artificial Tear
Number analyzed (Participants) | 113 | 114
Number of Patients
  Better | 8 | 7
  No Change | 104 | 107
  Worse | 1 | 0

5. Secondary Outcome: Change From Baseline of the Worse Eye in Corneal Topography as Measured by Pentacam at Day 90
Description: Change from Baseline in corneal topography of the worse eye as measured using a Pentacam system which calculates a number. Corneal topography is a non-invasive medical imaging technique for mapping the surface of the eye. The Pentacam system measures the pupil and anterior segment (the front part of the eye) which provides a range from 10 (best) to 60 (worst). A negative number change from baseline indicates an improvement.
Time Frame: Baseline, Day 90
Population: Intent-to-Treat population defined as all patients who started the study and were randomized
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Carboxymethylcellulose and Glycerin Based Artificial Tear | Carboxymethylcellulose Based Artificial Tear
Number analyzed (Participants) | 114 | 114
Units on a scale
  Baseline | 31.95 (11.941) | 32.32 (15.347)
  Change from Baseline at Day 90 | -2.12 (6.321) | -2.24 (6.267)

6. Secondary Outcome: Change From Baseline of the Worse Eye in Corneal Topography Measured by Humphrey Atlas at Day 90
Description: Change from Baseline in corneal topography of the worse eye as measured by a Humphrey Atlas system which calculates a number. Corneal topography is anon-invasive medical imaging technique for mapping the surface curvature of the cornea (the outer structure of the eye). The higher the number the more irregular the cornea. A Humphrey Atlas system detects irregular conditions in the cornea with a range from 0 = best to 2.5 = worst. A negative number change from baseline indicates an improvement.
Time Frame: Baseline, Day 90
Population: Intent-to-Treat population defined as all patients who started the study and were randomized
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Carboxymethylcellulose and Glycerin Based Artificial Tear | Carboxymethylcellulose Based Artificial Tear
Number analyzed (Participants) | 114 | 114
Units on a scale
  Baseline | 1.32 (0.855) | 1.25 (0.456)
  Change from Baseline at Day 90 | -0.49 (0.899) | -0.26 (0.396)

7. Secondary Outcome: Change From Baseline of Total Higher Order Aberration (HOA) of the Worse Eye at Day 90
Description: Change from Baseline in total HOA of the worse eye. The total HOA number is measured using a machine that calculates and detects changes in the cornea which could occur post Lasik surgery. A negative number change from baseline indicates an improvement.
Time Frame: Baseline, Day 90
Population: Intent-to-Treat population defined as all patients who started the study and were randomized
Measure: Mean (Standard Deviation); unit: Microns
Arm/Group | Carboxymethylcellulose and Glycerin Based Artificial Tear | Carboxymethylcellulose Based Artificial Tear
Number analyzed (Participants) | 114 | 114
Microns
  Baseline | 0.521 (0.1842) | 0.520 (0.1845)
  Change from Baseline at Day 90 | -0.058 (0.1509) | -0.047 (0.1452)

8. Secondary Outcome: Change From Baseline of the Worse Eye in Schirmer's Test at Day 90
Description: Change from baseline in Schirmer's Test results at Day 90 in the worse eye. The Schirmer's Test measures the rate of the secretion of tears produced by the eye over 5 minutes. The results indicate the presence of dry eye (Normal = greater than or equal to 15 millimeters (mm) of tears, Dry Eye = less than 15 mm of tears). The smaller the number, the more severe the dry eye.
Time Frame: Baseline, Day 90
Population: Intent-to-Treat population defined as all patients who started the study and were randomized
Measure: Mean (Standard Deviation); unit: Millimeters of Tears
Arm/Group | Carboxymethylcellulose and Glycerin Based Artificial Tear | Carboxymethylcellulose Based Artificial Tear
Number analyzed (Participants) | 114 | 114
Millimeters of Tears
  Baseline | 16.3 (8.40) | 13.5 (6.30)
  Change from Baseline at Day 90 | -0.3 (8.75) | 1.7 (9.59)

9. Secondary Outcome: Change From Baseline of the Worse Eye in Corneal Staining With Fluorescein at Day 90
Description: Change from Baseline in corneal staining of the worse eye at Day 90. Sum of corneal staining over 5 zones; each zone was measured on a modified Oxford Scheme (0 = no staining and 5 = severe staining), for a minimum score of 0 and a maximum score of 25. The higher the grade score, the worse the dry eye condition. A negative change from baseline represents a decrease in corneal staining (improvement).
Time Frame: Baseline, Day 90
Population: Intent to Treat population defined as all patients who started the study and were randomized
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Carboxymethylcellulose and Glycerin Based Artificial Tear | Carboxymethylcellulose Based Artificial Tear
Number analyzed (Participants) | 114 | 114
Scores on a Scale
  Baseline | 0.5 (1.13) | 0.5 (1.12)
  Change from Baseline at Day 90 | 0.0 (1.12) | 0.0 (1.47)

10. Secondary Outcome: Change From Baseline of the Worse Eye in Conjunctival Staining With Lissamine Green at Day 90
Description: Change from Baseline in conjunctival staining of the worse eye using Lissamine Green staining procedure. Sum of conjunctival staining over 6 zones; each zone was measured on a modified Oxford Scheme (0 = no staining and 5 = severe staining), with a minimum score of 0 and a maximum score of 30. The higher the grade score, the worse dry eye condition. A negative number change from baseline represents a decrease in corneal staining (improvement).
Time Frame: Baseline, Day 90
Population: Intent-to-Treat population defined as all patients who started the study and were randomized
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Carboxymethylcellulose and Glycerin Based Artificial Tear | Carboxymethylcellulose Based Artificial Tear
Number analyzed (Participants) | 114 | 114
Scores on a Scale
  Baseline | 1.0 (1.98) | 0.8 (1.32)
  Change from Baseline at Day 90 | 0.0 (1.65) | -0.3 (1.24)

11. Secondary Outcome: Change From Baseline of the Worse Eye in Tear Break-Up Time (TBUT) at Day 90
Description: Change from Baseline in TBUT of the worse eye at Day 90. TBUT is the time required for dry spots to appear on the surface of the eye after blinking. The longer it takes, the more stable the tear film. A short TBUT is a sign of poor tear film. A positive number change from baseline indicates an increase in TBUT (improvement).
Time Frame: Baseline, Day 90
Population: Intent-to-Treat population defined as all patients who started the study and were randomized
Measure: Mean (Standard Deviation); unit: Number of seconds
Arm/Group | Carboxymethylcellulose and Glycerin Based Artificial Tear | Carboxymethylcellulose Based Artificial Tear
Number analyzed (Participants) | 114 | 114
Number of seconds
  Baseline | 13.66 (6.133) | 13.25 (5.250)
  Change from Baseline at Day 90 | -0.92 (6.013) | -0.87 (12.924)

12. Other Pre Specified Outcome: Number of Patients Prescribed to Each Dosing Regimen at Day 14 and Day 60
Description: Number of patients prescribed to each dosing regimen at Day 14 and Day 60. At each visit from Day 14 (the first post-operative visit) to Day 60, patients were prescribed to 1 to 4 dosing regimens based on the investigator's clinical evaluation. Dosing schedule options were: At least every 2 hours while awake, 6 to 8 times per day, 3 to 5 times per day, at 1 to 2 times per day.
Time Frame: Day 14, Day 60
Population: Intent to Treat includes all patients that started the study and were randomized. Only those patients who were prescribed a dosing regimen at Day 14 to Day 60 visits were analyzed. The is indicated in parenthesis as (number of patients in arm 1 who were prescribed/number of patients in arm 2 who were prescribed).
Measure: Number; unit: Number of patients
Arm/Group | Carboxymethylcellulose and Glycerin Based Artificial Tear | Carboxymethylcellulose Based Artificial Tear
Number analyzed (Participants) | 114 | 114
Number of patients
  Day 14: at least every 2 hrs (113/110) | 20 | 22
  Day 14: 6-8 times a day (113/110) | 30 | 30
  Day 14: 3-5 times a day (113/110) | 58 | 54
  Day 14: 1-2 times a day (113/110) | 5 | 4
  Day 60: at least every 2 hrs (109/107) | 4 | 3
  Day 60: 6-8 times a day (109/107) | 12 | 14
  Day 60: 3-5 times a day (109/107) | 62 | 60
  Day 60: 1-2 times a day (109/107) | 31 | 30

13. Secondary Outcome: Change From Baseline in Study Product Usage at Day 90
Description: Change from baseline in the study product usage (average number of uses per day) at Day 90. A negative number change from baseline indicates a reduction in eye drop usage (improvement).
Time Frame: Baseline, Day 90
Population: Intent-to-Treat includes all patients that started the study and were randomized. Only those patients who reported actual eye drop use at Baseline and on Day 90 were analyzed. This is indicated in parenthesis as (number of patients in arm 1 who reported eye drop use/number of patients in arm 2 who reported eye drop use).
Measure: Mean (Standard Deviation); unit: Number of study product uses per day
Arm/Group | Carboxymethylcellulose and Glycerin Based Artificial Tear | Carboxymethylcellulose Based Artificial Tear
Number analyzed (Participants) | 114 | 114
Number of study product uses per day
  Baseline (108/108) | 7.9 (3.16) | 7.9 (4.89)
  Change from Baseline at Day 90 (108/105) | -4.9 (3.38) | -4.5 (5.97)

ADVERSE EVENTS:
Arm/Group | Carboxymethylcellulose and Glycerin Based Artificial Tear | Carboxymethylcellulose Based Artificial Tear
Serious Adverse Events (participants affected / at risk) | 0/114 | 0/114
Other Adverse Events (participants affected / at risk) | 88/114 | 82/114
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Carboxymethylcellulose and Glycerin Based Artificial Tear (N=114) | Carboxymethylcellulose Based Artificial Tear (N=114)
Punctate Keratitis (Eye disorders) | 21 | 22
Halo Vision (Eye disorders) | 10 | 9
Dry Eye (Eye disorders) | 10 | 8
Glare (Eye disorders) | 8 | 7
Conjucntival Haemorrhage (Eye disorders) | 8 | 6
Nasopharyngitis (Infections and infestations) | 8 | 6
Eye Operation Complications (Injury, poisoning and procedural complications) | 7 | 5
Foreign Body Sensation in Eyes (Eye disorders) | 6 | 6
Photophobia (Eye disorders) | 5 | 7
Ocular discomfort (Eye disorders) | 5 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.